CLINICAL TRIAL: NCT05442333
Title: Adjuvant Versus Neo-adjuvant Radiotherapy in Patients With Resectable Soft Tissue Sarcoma in Extremities : Wound Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ziad Khaled Abdullah Abdul Qader, orthopedic oncology department assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ziad khaled
Record Dates: First submitted 2022-04-15; First posted 2022-07-05 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Resectable Soft Tissue Sarcoma; Extremities; Radiotherapy Wound Complications

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative radiotherapy (Active Comparator): The patients which will receive preoperative radiotherapy
  Interventions: Procedure: surgical resection with safety margin
- postoperative radiotherapy (Active Comparator): The patients which will receive postoperative radiotherapy
  Interventions: Procedure: surgical resection with safety margin

INTERVENTIONS:
Procedure: surgical resection with safety margin — • The patients with preoperative radiotherapy:
  1. will be assessed 3 weeks post radiation regarding wound signs of infection (redness, hotness or discharge).
  2. 6 weeks post radiation for wound dehiscence
  3. 3 months post radiation for local swelling or recurrence
  4. 6 months post radiation for local recurrence, joint stiffness or pathological fractures.
  The patients with postoperative radiotherapy:
  1. will be assessed 3 weeks post radiation regarding wound signs of infection (redness, hotness or discharge).
  2. 6 weeks post radiation for wound dehiscence
  3. 3 months post radiation for local swelling or recurrence
  4. 6 months post radiation for local recurrence, joint stiffness or pathological fractures.
  Other Names: pre operative radiotherapy; post operative radiotherapy

SUMMARY:
Extremity soft tissue sarcomas (ESTS)s are rare mesenchymal cancers that considered a challenge for orthopaedic surgeons. Soft tissue sarcomas (STS) comprise less than 1% of malignant cancers, commonly occur in the proximal extremities and trunk. Limb-sparing surgery mostly are targeted in most of the patients, so adjuvant or neoadjuvant radiotherapy is usually added. Preoperative radiotherapy (neoadjuvant) or postoperative radiotherapy (adjuvant) offers local control and survival rates, but the local complications are controversial. However, different retrospective studies had shown that preoperative radiotherapy cause higher wound complication rate, while both preoperative and postoperative radiotherapy had the same results regarding local recurrence

DETAILED DESCRIPTION:
Study Tools :The patients will be managed as follows:

Primary (Preoperative) Diagnosis and Evaluation

Clinical Evaluation. History. General examination. Local examination.

Radiological Evaluation:

Plain X-ray for the affected limb to determine presence of any bone affection or invasion.

Preoperative MRI scan to determine the extent of soft tissue, bone and neurovascular bundle invasion.

Preoperative bone scan to determine skeletal metastatic load.

Perioperative protocol:

Preoperative radiotherapy 3-6 weeks before surgical excision. Postoperative radiotherapy 3- 6 weeks or more after surgical excision Tissue diagnosis will be obtained.

Operative management:

Surgical excision of whole tumour with wide safety margin.

Data collection:

Patient demographics (age, sex). Activity level Primary sarcoma type Patient comorbidities Timing of Preoperative radiotherapy if present. Timing of Postoperative radiotherapy if present. Time from diagnosis to surgery. recurrence Operative time (minutes) measured from skin incision to wound closure. Follow up regarding wound complications, local recurrence or infection. local recurrence will be followed up till the end of the study

Follow up strategy:

The patients with preoperative radiotherapy:

will be assessed 2 weeks postoperative regarding wound signs of infection (redness, hotness or discharge).

1 month postoperatively for wound complete closure and exclude signs of infection.

3 months postoperatively for wound dehiscence, swelling or local recurrence. 6 months postoperatively for local recurrence, pathological fractures or joint stiffness

The patients with postoperative radiotherapy:

will be assessed 3 weeks post radiation regarding wound signs of infection (redness, hotness or discharge).

6 weeks post radiation for wound dehiscence 3 months post radiation for local swelling or recurrence 6 months post radiation for local recurrence, joint stiffness or pathological fractures.

Statistical Analysis: Statistical package for social science (SPSS 15.0.1 for windows ; 〖SPSS Inc,Chicago,IL,2001). Data will be presented as Mean and Standard deviation ( +/-SD) for quantitative parametric data , and Median and Interquartile range for quantitative non parametric data. Frequency and percentage will be used for presenting qualitative data. Suitable analysis will be done according to the type of data obtained. P<0.05 will be considered significant.

Statistical Package: data entry and statistical analysis of the collected data will be performed using reliable software program.

ELIGIBILITY:
Inclusion Criteria:

* Sex: both sexes.
* Lesion: any soft tissue sarcoma in upper or lower limbs (synovial sarcoma, liposarcoma, fibrosarcoma and others)
* age more than 16 years old

Exclusion Criteria:

* Irresectable ESTS
* Round cell ESTS
* recurrent ESTS
* patients who received local irradiation due to other causes

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
wound and local complications | 12 months

SECONDARY OUTCOMES:
recurrence rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months